CLINICAL TRIAL: NCT05206877
Title: Topical Insulin for Glaucoma and Optic Neuropathies
Brief Title: Topical Insulin for Glaucoma
Acronym: TING1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey L Goldberg, Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 63337
Record Dates: First submitted 2022-01-06; First posted 2022-01-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Low dose topical insulin (Experimental): Group 1; N=6: 100 U/ml; 4 units of insulin per application, 1 drop done in clinic daily for 5 days
  Interventions: Drug: Insulin, 4 units
- High dose topical insulin (Experimental): Group 2; N=6: 500 U/ml; 20 units of insulin per application, 1 drop done in clinic daily for 5 days
  Interventions: Drug: Insulin, 20 units
- Longer-term topical insulin (Experimental): Group 3 randomized; N=20: 10 subjects will receive the highest tolerated dose (e.g. from group 1 or group 2), 1 drop per day at home for 1 month, full testing pre- and post-treatment, and 10 subjects will receive 1/5 of the highest tolerated dose (either the lower dose, or if needed will dilute) 1 drop per day at home for 1 month, full testing pre- and post-treatment.
  Interventions: Drug: Insulin, 4 units; Drug: Insulin, 20 units
- Low-Dose Insulin twice Daily (Experimental): Group 4. N=5. 1 drop of 100U/mL insulin administered twice daily for 5 days.
  Interventions: Drug: insulin, 4 units twice daily
- High-Dose Insulin twice Daily (Experimental): Group 5. N=5. 1 drop of 500U/mL insulin administered twice daily for 5 days.
  Interventions: Drug: insulin, 20 units twice daily
- Low-Dose Insulin three times daily (Experimental): Group 6. N=5. 1 drop of 100U/mL insulin administered three times daily for 5 days.
  Interventions: Drug: insulin, 4 units three times daily
- High-Dose Insulin three times daily (Experimental): Group 7. N=5. 1 drop of 500U/mL insulin administered three times daily for 5 days.
  Interventions: Drug: insulin, 20 units three times daily

INTERVENTIONS:
Drug: Insulin, 4 units — Topical insulin 100 U/ml, 1 drop per day
  Arms: Longer-term topical insulin; Low dose topical insulin
Drug: Insulin, 20 units — Topical insulin 500 U/ml, 1 drop per day
  Arms: High dose topical insulin; Longer-term topical insulin
Drug: insulin, 4 units twice daily — 1 drop of low dose insulin twice daily.
  Arms: Low-Dose Insulin twice Daily
Drug: insulin, 20 units twice daily — 1 drop of high dose insulin twice daily
  Arms: High-Dose Insulin twice Daily
Drug: insulin, 4 units three times daily — 1 drop of low dose insulin three times daily.
  Arms: Low-Dose Insulin three times daily
Drug: insulin, 20 units three times daily — 1 drop of high dose insulin three times daily.
  Arms: High-Dose Insulin three times daily

SUMMARY:
The purpose of this Phase 1 trial is to determine the safety over 1-2 months of topic sterile human recombinant insulin on subjects with optic neuropathies (glaucoma, ischecmic optic neuropathy, and optic disc drusen).

ELIGIBILITY:
Inclusion Criteria:

* Capable to provide informed consent
* Diagnosis of optic neuropathy either glaucoma or NAION or optic disc drusen.
* Only one eye per patient will be selected as the study eye - if both eyes meet the inclusion criteria, the eye with the worse acuity and /or visual field will be selected. The contralateral eye will be left untouched.

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Presence of any ocular pathologies other than glaucoma that contributes to the severe vision loss (retinopathy / maculopathy, severe uveitis, keratopathy, etc.)
* Diagnosis of glucose intolerance, type 1 or 2 diabetes mellitus
* Inability to perform reliable visual field
* Unable to provide informed consent
* Unable to complete the tests and follow-ups required by the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | During treatment period, difference from baseline to post-treatment up to 2 months
  determine the safety of topical sterile human insulin in patients with optic neuropathies. AEs and SAEs will be monitored and recorded through the duration of the study.

SECONDARY OUTCOMES:
Change in retinal thickness measured in microns by spectral domain optical coherence tomography (sdOCT) | During treatment period, difference from baseline to post-treatment up to 2 months
  The change in retinal thickness as measured by spectral domain optical coherence tomography (sdOCT)
The change in visual field as measured by mean deviation | During treatment period, difference from baseline to post-treatment up to 2 months
  The change in visual field as measured by mean deviation on Zeiss Humphrey Visual Field testing

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Goldberg, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share individual participant data